CLINICAL TRIAL: NCT01916421
Title: The Cellularity Yield of Three Different 22-gauge Endoscopic Ultrasound Fine Needle Aspiration Needles
Brief Title: The Cellularity Yield of Three Different 22-gauge FNA Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Mohamed O Othman, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E12097
Record Dates: First submitted 2013-06-23; First posted 2013-08-05 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic or Peripancreatic Lesions; Lesions in the Esophagus, Stomach, Duodenum or Rectum; Mediastinal ( Chest) Masses; Enlarged Lymph Nodes
Keywords: Pancreatic adenocarcinoma; lymphadenopathy; Endoscopic ultrasound
MeSH Terms: conditions — Lymphadenopathy | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EZ Shot (Active Comparator)
  Interventions: Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA)
- Expect™ (Active Comparator)
  Interventions: Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA)
- EchoTip® Ultra (Active Comparator)
  Interventions: Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA)

INTERVENTIONS:
Procedure: Endoscopic Ultrasound Fine Needle Aspiration (EUS-FNA)

SUMMARY:
Obtaining a sample from a lesion in the gastrointestinal tract by endoscopic ultrasound (a flexible tube with a camera and small ultrasound machine at its end )requires the use of a needle for taking the sample from the lesion or what we call "Fine needle aspiration (FNA)". Currently, FNA is done by three commercially available needles. These needles are used routinely in our institution for FNA. The data regarding the safety and the successfulness of any of these needles are lacking. We sought to compare all three commercially available needles in a prospective manner.

DETAILED DESCRIPTION:
The following are being done only for research purposes; prior to performing the FNA, The patient will be randomized to one of the three commercially available FNA needles. At this time, all needles are considered equivalent and there is no medical necessity to pick one over another. The sample obtained by the needle will be assigned a quality score based on certain parameters of the sample such as the abundance of diagnostic cells and the presence of blood. We are going to collect certain information about your procedure such as the complications of the procedure, number of needle passes and final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18-88) who are undergoing EUS FNA of pancreatic or peripancreatic lesions
2. Adult patients (18-88) who are undergoing EUS FNA of submucosal masses in the esophagus, stomach, duodenum or rectum
3. Adult patients (18-88) who are undergoing EUS FNA of mediastinal masses.
4. Adult patients (18-88) who are undergoing EUS FNA of enlarged lymph nodes

Exclusion Criteria:

1. Patients younger than 18 yrs old or older than 88 yrs.
2. Pregnant patients

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
1. Compare the overall diagnostic accuracy of the three commercially available 22 gauge EUS needles | 2 days after the procedure
  Cellularity score will be assessed by the cytopathologist using the scoring system from 0 to 10 score. This scoring system evaluate the amount of blood, malignant cells and contaminant cells. The system is a modified form Mair et al study. " Mair S, Dunbar F, Becker PJ, Du Plessis W. Fine needle cytology--is aspiration suction necessary? A study of 100 masses in various sites. Acta cytologica 1989;33:809-13."

SECONDARY OUTCOMES:
Compare the complication rate between the three commercially available 22 gauge EUS needles. | up to 1 month after the procedure
  The patient will be contacted after the procedure by one week to review any procedure complications. The patient's medical records may be reviewed for up to 6 months after the procedure to review the surgical resection results or the long-term follow-up results. If the patient receives his further care in another hospital, the patient will be contacted by phone for follow-up for a maximum period of 6 months.
Compare the number of FNA needles passes required to reach the diagnosis. | During the procedure ( 30 -45 minutes)
  The number of passes required to reach the diagnosis
Compare the technical success of the three commercially available 22 gauge EUS needles | During the procedure ( 30-45 minutes)
  The ability of the needle to perform the intended purpose of the procedure ( reach the lesion and obtain sufficient tissues)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed O Othman, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Sciences Center at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No